CLINICAL TRIAL: NCT06245356
Title: TRIFLUOX-DP: Safety of Trifluridine/Tipiracil as Replacement of Fluoropyrimidines (5-fluorouracil and Capecitabine) Based Chemotherapy as First Line Metastatic Colorectal or Gastroesophageal Cancer Regimens in Patients With Dihydropyrimidine Dehydrogenase Deficiency: a Phase II Trial
Brief Title: Safety of Trifluridine/Tipiracil in Patients With Dihydropyrimidine Dehydrogenase Deficiency Diagnosed With Metastatic Colorectal or Gastroesophageal Cancer
Acronym: TRIFLUOX-DP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 91 - UCGI 46
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Gastroesophageal Adenocarcinoma; DPD Deficiency
Keywords: Metastatic colorectal cancer; Metastatic Gastroesophageal Adenocarcinoma; DPD Deficiency; Trifluridine/Tipiracil
MeSH Terms: conditions — Colorectal Neoplasms; Dihydropyrimidine Dehydrogenase Deficiency | interventions — trifluridine tipiracil drug combination; Oxaliplatin; Panitumumab; Bevacizumab; Trastuzumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colorectal adenocarcinoma (Other): Trifluridine/tipiracil in association with oxaliplatin with or without:
  * Panitumumab in RAS wild type tumors
  * Bevacizumab in RAS wild type of right colon or RAS mutated tumors
  Interventions: Drug: Lonsurf; Drug: Oxaliplatin; Drug: Panitumumab; Drug: Bevacizumab
- Gastroesophageal adenocarcinoma (Other): Trifluridine/tipiracil in association with oxaliplatin with or without:
  * Trastuzumab in HER2-positive tumors (3+ IHC or 2+/FISH+)
  * Nivolumab if CPS≥5 and HER2-negative tumors
  Interventions: Drug: Lonsurf; Drug: Oxaliplatin; Drug: Trastuzumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Lonsurf — Trifluridine/tipiracil orally 35 mg/m²/dose (D1-D5 twice daily, D1=D15)
Drug: Oxaliplatin — Oxaliplatin intravenous injection 85 mg/m² every 2 weeks (D1=D15)
Drug: Panitumumab — Panitumumab intravenous injection 6 mg/kg (D1=D15)
  Arms: Colorectal adenocarcinoma
Drug: Bevacizumab — Bevacizumab intravenous injection 5 mg/kg (D1=D15)
  Arms: Colorectal adenocarcinoma
Drug: Trastuzumab — Trastuzumab intravenous injection 4 mg/kg (D1=D15)
  Arms: Gastroesophageal adenocarcinoma
Drug: Nivolumab — Nivolumab intravenous injection 240 mg (D1=D15)
  Arms: Gastroesophageal adenocarcinoma

SUMMARY:
The goal of this clinical trial is to test the safety of the trifluridine/tipiracil as replacement of fluoropyrimidines based chemotherapy as first line metastatic colorectal or gastroesophageal cancer regimens in patients with dihydropyrimidine dehydrogenase (DPD) deficiency.

The main questions it aims to answer are:

* Is this alternative chemotherapy option a better option in term of safety for this type of patients?
* Does the combination of treatments improves the overall safety?
* Does the combination of treatments improves the progression-free survival, overall survival, objective response rate and disease control rate?
* Does the combination of treatment have an effect on quality of life?

Participants will:

* Receive the trifluridine/tipiracil with oxaliplatin every 14 days, associated with:

  * Panitumumab or bevacizumab for colorectal adenocarcinomas
  * Nivolumab or trastuzumab for gastroesophageal adenocarcinomas.
* Have a CT-Scan every 2 months until disease progression
* Complete Health-related quality of life questionnaire every 2 months for a maximum of 6 months
* Participate to the optional translational research: Blood samples fo DPYD genotyping and pharmacokinetic analysis

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed and dated a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
2. Histological or cytological documentation of adenocarcinoma of the colon or rectum or gastroesophageal cancer (lower oesophagus, gastroesophageal junction and gastric)
3. Synchronous or metachronous metastatic colorectal or gastroesophageal cancer
4. Presence of at least one measurable lesion according to RECIST v1.1
5. No prior therapy for metastatic disease
6. known DPD deficiency defined as plasma uracil concentration≥16 ng/ml For plasma uracil concentration [16-20[ ng/ml, plasma uracil dosage must be repeated in the 7 days to confirm that plasma uracil concentration ≥16 ng/ml. If the second result is different (i.e; uracil concentration <16 ng/ml), keep the favourable result, and do not include the patient if only the first plasma uracil concentration≥16 ng/ml.
7. Age ≥18 years
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
9. Adequate bone marrow, renal and liver functions as evidenced by the following laboratory requirements within 7 days prior to study treatment initiation:

   1. Absolute neutrophil count (ANC) ≥ 1,500/ mm³ without biologic response modifiers such as granulocyte colony-stimulating factor (G-CSF), within 21 days before the start of study treatment
   2. Platelet count ≥100,000/mm³, without platelet transfusion within 21 days before the start of study treatment
   3. Hemoglobin (Hb) ≥9 g/dL, without blood transfusion or erythropoietin within 21 days before the start of study treatment
   4. Serum creatinine ≤1.5 x upper limit of normal (ULN)
   5. Glomerular filtration rate as assessed by the estimated glomerular filtration rate (eGFR) ≥50 mL/min per 1.73 m² calculated by the Modification of Diet in Renal Disease (MDRD) abbreviated formula
   6. Total bilirubin ≤ 1.5 x ULN
   7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement of their cancer)
   8. Alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 5.0 x ULN for patients with liver involvement for their cancer and/or bone metastases)
   9. International normalized ratio (INR) ≤1.5 or prothrombin time (PT) ≤1.5 x ULN Note: Patients on stable dose (dose has not been changed in at least 28 days) of anticoagulation therapy will be allowed to participate if they have no sign of bleeding or clotting and INR / PT and PTT / aPTT test results are compatible with the acceptable benefit-risk ratio at the investigator's discretion. In such case, limits as noted would not apply
10. For women of reproductive potential, negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test obtained within 7 days before the start of study treatment. Women not of reproductive potential are female patients who are postmenopausal or permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy)
11. For women of childbearing potential and men, agreement to use an adequate contraception for the duration of study participation and up to 7 months following completion of therapy.
12. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
13. Affiliation to the Social Security System (or equivalent).

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from colorectal or gastroesophageal cancer within 5 years prior to study inclusion, except for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non invasive tumor), Tis (carcinoma in situ) and T1 (lamina propria invasion)]
2. Radiotherapy within 28 days prior to first dose of treatment
3. Active cardiac disease including any of the following:

   1. Symptomatic Congestive heart failure ≥New York Heart Association (NYHA) class 3 or 4
   2. Severe Unstable angina (angina symptoms at rest)
   3. Myocardial infarction less than 12 months before first dose of treatment
4. Uncontrolled hypertension (Systolic blood pressure ≥140 mmHg or diastolic pressure ≥ 90 mmHg) despite optimal medical management.
5. Ongoing infection ≥Grade 2 (NCI CTCAE v.5.0)
6. Known history of human immunodeficiency virus (HIV) infection
7. Chronic hepatitis B or C infection (if hepatitis status cannot be obtained from medical records, re-testing is required)
8. Seizure disorder requiring medication
9. Symptomatic metastatic brain or meningeal tumours
10. History of organ allograft
11. Known hypersensitivity to any of the study drugs, study drug classes, or any constituent of the products
12. In case of planned treatment with oxaliplatin: Peripheral neuropathy >Grade 1 (NCI CTCAE v.5.0)
13. In case of planned treatment with bevacizumab: Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to first dose of treatment
14. In case of planned treatment with bevacizumab: Evidence or history of any bleeding diathesis, irrespective of severity. Any hemorrhage or bleeding event ≥CTCAE v 5.0 Grade 3 within 4 weeks prior to the start of study medication
15. In case of planned treatment with trastuzumab or panitumumab or bevacizumab: Interstitial lung disease with ongoing signs and symptoms
16. Inability to swallow oral medication
17. Any uncontrolled malabsorption condition
18. Pregnant or breast-feeding subjects. Women of childbearing potential must have a serum pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of study drug
19. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, substance abuse, medical or psychological reasons, or any condition that, in the opinion of the investigator, would interfere with the patient's participation in the study or evaluation of study treatment or interpretation of patient safety or study results
20. Participation in another clinical study with an investigational product during the last 30 days before inclusion
21. Patients who might be interconnected with or dependent on the sponsor site or the investigator
22. Persons deprived of their liberty or under protective custody or guardianship, or legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-10-22 (Estimated); Study Completion 2028-10-21 (Estimated)

PRIMARY OUTCOMES:
Treatment specific safety | 1 month
  The percentage of patients without specific toxicities defined as grade 3-4-5 digestive toxicities (diarrhoea and/or stomatitis) and grade 4-5 neutropenia or febrile neutropenia over the first 2 cycles of first-line metastatic treatment.
  Toxicities will be graded using the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5), widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.

SECONDARY OUTCOMES:
Overall Safety | Throughout study completion, up to 2 years
  All types of toxicities occuring during the study. The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Compliance with study treatment | 1 month
  Patients will record Trifluridine/tipiracil intake within a leaflet every day. Investigators will collect this data at every on site visit during the first 2 cycles (before Cycle 3).
Progression Free Survival | From baseline until disease progression or death, up to 2 years
  The progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.
Overall Survival | From baseline until disease progression or death, up to 2 years
  The overall survival is the length of time from baseline that patients enrolled in the study are still alive.
Objective response rate | From baseline until disease progression, up to 2 years
  The objective response rate is defined as the percentage of patients with a complete response (CR) or a partial response (PR) for a given treatment.
Disease control rate | From baseline until disease progression, up to 2 years
  The disease control rate is defined as the percentage of patients with a CR, a PR or stable disease for a given treatment.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, 2 months, 4 months, and 6 months
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire - Oesophago-Gastric (QLQ-OG25) | At baseline, 2 months, 4 months, and 6 months
  This EORTC oesophago-gastric cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-OG25 contains 25 items organized into six scales: dysphagia (three items), eating restrictions (four items), reflux (two items), odynophagia (two items), pain and discomfort (two items) and anxiety (two items), and ten single items: eating in front of others, dry mouth, trouble with taste, body image, trouble swallowing saliva, choked when swallowing, trouble with coughing, trouble talking, weight loss and hair loss. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Quality of life questionnaire - Colorectal (QLQ-CR29) | At baseline, 2 months, 4 months, and 6 months
  This EORTC colorectal cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-CR29 has 5 functional and 18 symptom scales. It contains 29 items organized into four subscales: urinary frequency (two items), blood and mucus in stool (two items), stool frequency (two items), and body image (three items), and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest, impotence, sexual interest, and dyspareunia). All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle SAMALIN, MD, Principal Investigator — Institut du Cancer de Montepllier
Locations (21):
- France (21):
  - CHU Amiens, Amiens
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut du Cancer d'Avignon, Avignon
  - CHU Jean Minjoz, Besançon
  - Centre Hospitalier de Cholet, Cholet
  - Centre Georges François Leclerc, Dijon
  - Hôpital Privé Jean Mermoz, Lyon
  - Institut Régional du Cancer de Montpellier - ICM Val d'Aurelle, Montpellier
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital des Diaconesses Croix Saint Simon, Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHU de REIMS, Reims
  - Institut Godinot, Reims
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - CHU Saint-Etienne, Saint-Priest-en-Jarez
  - CH de Saint-Malo, St-Malo
  - Hôpital Nord Franche-Comté / Site du Mittan, Trévenans
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy